CLINICAL TRIAL: NCT00484185
Title: Post Marketing Surveillance To Observe Safety And Efficacy Of BeneFIX In Patients With Hemophilia B
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 3090X1-4403; B1821005
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Results first posted 2013-08-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-05

CONDITIONS: Hemophilia B
Keywords: Hemophilia B; BeneFIX; Safety; Efficacy
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Drug: BeneFIX (coagulation factor IX (recombinant))

INTERVENTIONS:
Drug: BeneFIX (coagulation factor IX (recombinant)) — BeneFIX will be administered according to physician's discretion.

SUMMARY:
To provide safety and effectiveness information of BeneFIX during the post-marketing period as required by Korea FDA regulations, to identify any potential drug related treatment factors in Korean population including:

1) Unknown adverse reactions, especially serious adverse reactions; 2) Changes in the incidences of adverse reactions under the routine drug uses.

3) Factors that may affect the safety of the drug 4) Factors that may affect the effectiveness of the drug

DETAILED DESCRIPTION:
The patients who meet the inclusion criteria will be enrolled consecutively.

ELIGIBILITY:
Inclusion Criteria:

* Patients or legally authorized representatives of pediatric patients agree to provide written informed consent form (data privacy statement).
* Pediatric and adult patients who have been treated with original or reformulated BeneFIX for hemophilia B (congenital factor IX deficiency or Christmas disease) from first approved date by KFDA, or who are planned to be newly prescribed BeneFIX (for example, patients switching from pdFIX to BeneFIX).

Exclusion Criteria:

* Patients with a known history of hypersensitivity to original or reformulated BeneFIX or any component of the product.
* Patients with a known history of hypersensitivity to hamster protein.
* Patients participating in an interventional trial of any investigational drug or device.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hemophilia B (congenital factor IX deficiency or Christmas disease).
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2007-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Seoul, South Korea

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3090X1-4403&StudyName=Post%20Marketing%20Surveillance%20To%20Observe%20Safety%20and%20Efficacy%20Of%20BeneFIX%20In%20Patients%20With%20Hemophilia%20B

RESULTS

PARTICIPANT FLOW:
Groups:
- BeneFIX: Participants who received original or reformulated BeneFIX (recombinant coagulation factor IX) infusion intravenously as indicated according to the approved local product document, dosage solely adjusted as per physician's discretion, were observed for a period of 6 months.
Period: Overall Study
Arm/Group | BeneFIX
Started | 183
Treated | 178
Completed | 112
Not Completed | 71
Not completed — Lost to Follow-up | 44
Not completed — Other | 20
Not completed — Randomized but not treated | 5
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | BeneFIX
Number analyzed (Participants) | 178
Age Continuous [Mean (Standard Deviation); unit: years] | 25.1 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 177

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) According to Baseline Characteristics
Description: AE: any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. AE assessed by baseline characteristics (chr) included age, gender, pediatric/geriatric status, liver disorder, BeneFIX treatment (previously/newly), factor nine (FIX) gene mutation, prior exposure to plasma-derived FIX products, prior FIX regimen(s) utilized, personal history of FIX inhibitor, family history of hemophilia B, severity of bleeding, medical history, concomitant medication and therapy.
Time Frame: Baseline up to 6 months
Population: Safety analysis set included all participants who received at least 1 dose of study medication including dropouts due to AEs.
Measure: Number; unit: participants
Arm/Group | BeneFIX
Number analyzed (Participants) | 178
participants
  Age: Less than (<) 10 years | 0
  Age: 10 to 19 years | 1
  Age: 20 to 29 years | 2
  Age: 30 to 39 years | 3
  Age: 40 to 49 years | 1
  Age: Greater than or equal (>=) to 50 years | 2
  Gender: Male | 9
  Gender: Female | 0
  Pediatric status: < 12 years | 0
  Pediatric status: >= 12 years | 9
  Geriatric status: < 65 years | 8
  Geriatric status: >= 65 years | 1
  Liver disorder: Yes | 2
  Liver disorder: No | 7
  BeneFIX treatment: New | 0
  BeneFIX treatment: Previous | 9
  Factor IX gene mutation: Yes | 0
  Factor IX gene mutation: No | 1
  Factor IX gene mutation: Unknown | 8
  Exposed to plasma-derived FIX products: Yes | 5
  Exposed to plasma-derived FIX products: No | 1
  Exposed to plasma-derived FIX products: Unknown | 3
  Prior FIX regimen: Yes | 8
  Prior FIX regimen: No | 1
  Personal history of FIX inhibitor: Yes | 1
  Personal history of FIX inhibitor: No | 8
  Family history of hemophilia B: Brother | 1
  Family history of hemophilia B: Other | 1
  Family history of hemophilia B: None | 6
  Family history of hemophilia B: Unknown | 1
  Severity: Mild | 0
  Severity: Moderate | 4
  Severity: Severe | 4
  Severity: Unknown | 1
  Medical history: Yes | 6
  Medical history: No | 3
  Concomitant medication: Yes | 5
  Concomitant medication: No | 4
  Concomitant therapy: Yes | 2
  Concomitant therapy: No | 7

2. Primary Outcome: Number of Participants With Adverse Events (AEs) According to Severity
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AE was assessed according to severity; mild (not causing any significant problem, dose adjustment not required), moderate (caused problem that does not interfere significantly with usual activities or the clinical status, dose adjustment needed due to adverse event) and severe (caused problem that interferes significantly with usual activities or the clinical status, study drug stopped due to adverse event).
Time Frame: Baseline up to 6 months
Population: Safety analysis set included all participants who received at least 1 dose of study medication including dropouts due to AEs. Same participant may be represented in more than 1 category.
Measure: Number; unit: participants
Arm/Group | BeneFIX
Number analyzed (Participants) | 178
participants
  Mild | 6
  Moderate | 2
  Severe | 4

3. Primary Outcome: Number of Participants With Action Taken in Response to Adverse Events (AEs)
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. After an onset of an AE, relevant actions were undertaken on the study drug or the participant. Actions related to study drug included: dosage reduced, dosage increased, stopped temporarily or permanently, no action taken; actions related to participants included: withdrawal from the study, concomitant medication, no action taken or any other as per physician's discretion.
Time Frame: Baseline up to 6 months
Population: Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis.
Arm/Group | BeneFIX
Number analyzed (Participants) | 0

4. Primary Outcome: Number of Participants With Adverse Events (AEs) According to Seriousness
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Seriousness of an AE was assessed under the criteria of serious adverse event (SAE). An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | BeneFIX
Number analyzed (Participants) | 178
participants
  SAEs | 4
  Non-SAEs | 5

5. Primary Outcome: Number of Participants With Outcome in Response to Adverse Events (AEs)
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Outcome of an AE was assessed based on response to a question 'Is the adverse event still present?' as 'yes', 'unknown' or 'no-resolved'.
Time Frame: Baseline up to 6 months
Population: as for outcome 3
Arm/Group | BeneFIX
Number analyzed (Participants) | 0

6. Primary Outcome: Number of Participants With Adverse Events (AEs) by Relationship
Description: AE: untoward medical occurrence in participant who received study drug without regard to causal relationship. All causalities and drug-related AEs reported. Drug-related AEs based on physician's discretion: certain (AE after drug intake, not explained by other drugs, reaction on drug cessation [DC], relapse on re-intake of drug), probable/likely (AE after drug intake, not explained by other drugs, reaction on DC, no information on re-intake), possible (AE after drug intake, explained by other drugs, no information on DC), unlikely (not related to drug intake time, explained by other drugs).
Time Frame: Baseline up to 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | BeneFIX
Number analyzed (Participants) | 178
participants
  AEs (all-causalities) | 9
  AEs (drug-related) | 1

7. Primary Outcome: Number of Participants With Unexpected Adverse Events (AEs)
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Unexpected AEs were those that were not included in precaution of local product document.
Time Frame: Baseline up to 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | BeneFIX
Number analyzed (Participants) | 178
participants | 0

8. Secondary Outcome: Mean Annualized Bleeding Rate (ABR)
Description: An annualized bleeding rate (ABR) was calculated as the number of bleeds requiring administration of BeneFIX (for on-demand therapy and surgery), divided by total period of bleeding multiplied by 365.25. Total period of bleeding is the number of days on treatment for prophylaxis purpose and on-demand therapy and surgery.
Time Frame: Baseline up to 6 months
Population: Efficacy analysis set included all participants who received at least 1 dose of study medication for the approved indications and were evaluated upon its related parameters at least once. Here 'N' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: bleeds per year
Arm/Group | BeneFIX
Number analyzed (Participants) | 135
bleeds per year | 84.25 (125.35)

9. Secondary Outcome: Number of Responses to On-demand Treatment With Study Medication
Description: Responses to on-demand treatment were rated by participant/caregiver or physician each time the drug was administered, on 4-point scale. Score 1=excellent (definite pain relief [PR] and improvement [imp] within 8 hours [h] of infusion [inf], no additional inf); score 2=good (definite PR and imp within 8h of inf, at least 1 additional inf for complete resolution [CR] of bleeding or starting after 8h of inf, no additional inf); score 3=moderate (probable or slight imp starting after 8h of inf, at least 1 additional inf for CR of bleeding); score 4=no imp at all, or condition worsens).
Time Frame: Baseline up to 6 months
Population: as for outcome 8
Measure: Number; unit: responses
Arm/Group | BeneFIX
Number analyzed (Participants) | 135
responses
  Excellent | 1145
  Good | 788
  Moderate | 65
  No response | 0

10. Secondary Outcome: Mean Number of Infusion of Study Medication
Description: Mean frequency of BeneFIX administration of each participant was calculated from number of BeneFIX infusions which each participant received for treatment of each new bleed. Mean frequency of BeneFIX administration for total participants was summarized.
Time Frame: Baseline up to 6 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: infusions
Arm/Group | BeneFIX
Number analyzed (Participants) | 135
infusions | 2.25 (4.33)

11. Secondary Outcome: Mean Number of Breakthrough Bleeds Within 48 Hours of Study Medication
Description: Mean frequency of breakthrough (spontaneous/non-traumatic) bleeds of each participant within 48 hours of a preventive/prophylaxis dose of BeneFIX was calculated from number of irregular bleeding which occurred in each participant. Mean frequency breakthrough bleeds for total participants within 48 hours of a preventive/prophylaxis dose of BeneFIX was summarized.
Time Frame: Baseline up to 6 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: breakthrough bleeds
Arm/Group | BeneFIX
Number analyzed (Participants) | 123
breakthrough bleeds | 0.27 (0.47)

12. Secondary Outcome: Average Infusion Dose of Study Medication
Description: Average of dose per infusion per kilogram (kg) body weight was reported for prophylaxis purpose or on-demand therapy and surgery.
Time Frame: Baseline up to 6 months
Population: Efficacy analysis set included all participants who received at least 1 dose of study medication for the approved indications and were evaluated upon its related parameters at least once. Here 'N' (number of participants analyzed)= participants evaluable for this measure and 'n' = participants evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: international unit/kilogram (IU/kg)
Arm/Group | BeneFIX
Number analyzed (Participants) | 135
international unit/kilogram (IU/kg)
  On-demand therapy and surgery: n= 135 | 38.79 (5.41)
  Prophylaxis purpose: n= 123 | 32.92 (10.43)

13. Secondary Outcome: Total Infusion of Study Medication
Description: Total dose of study drug infused was calculated over the study duration.
Time Frame: Baseline up to 6 months
Population: Efficacy analysis set included all participants who received at least 1 dose of study medication for the approved indications and were evaluated upon its related parameters at least once.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | BeneFIX
Number analyzed (Participants) | 178
IU | 50356.11 (42154.05)

14. Secondary Outcome: Percentage of Participants With Efficacy Evaluation
Description: The efficacy of study drug was rated as 'very effective', 'effective', 'slightly ineffective' and 'ineffective'.
Time Frame: Baseline up to 6 months
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | BeneFIX
Number analyzed (Participants) | 11
percentage of participants
  Very effective | 81.82
  Effective | 18.18
  Slightly ineffective | 0.00
  Ineffective | 0.00

15. Other Pre Specified Outcome: Duration of Adverse Events (AEs)
Description: Total time from onset of adverse event till the event is resolved. Duration of AE per event = AE stop date minus AE start date plus 1.
Time Frame: Baseline up to 6 months
Population: as for outcome 3
Arm/Group | BeneFIX
Number analyzed (Participants) | 0

16. Other Pre Specified Outcome: Number of Participants Who Discontinued the Study Due to Adverse Events (AEs)
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Number of participants who discontinued the study due to AEs was reported.
Time Frame: Baseline up to 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | BeneFIX
Number analyzed (Participants) | 178
participants | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | BeneFIX
Serious Adverse Events (participants affected / at risk) | 4/178
Other Adverse Events (participants affected / at risk) | 5/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BeneFIX (N=178)
Drug ineffective (General disorders) | 1
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BeneFIX (N=178)
Stomatitis (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.